CLINICAL TRIAL: NCT06034535
Title: CD62L Depleted Donor Lymphocyte Infusion With T Cell Depleted Haploidentical Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Cheuk Ka Leung Daniel, Consultant, Hong Kong Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKCH-REC-2022-002
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Hematopoietic Organs; Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): CD62L depleted donor lymphocyte infusion
  Interventions: Biological: CD62L depleted donor lymphocyte infusion

INTERVENTIONS:
Biological: CD62L depleted donor lymphocyte infusion — Intravenous infusion of CD62L depleted donor lymphocytes

SUMMARY:
In this clinical trial, the investigators aim to apply CD62L depleted donor lymphocyte infusion (DLI) together with in vitro T cell depleted haploidentical hematopoietic stem cell transplantation (HSCT) to treat patients with malignant or non-malignant disease in need of HSCT. The investigators shall evaluate the graft failure-free, graft-versus-host disease (GVHD)-free survival at one year, frequency of adverse events and post-transplant complications, and immunoreconstitution.

DETAILED DESCRIPTION:
The peripheral stem cell harvest product from the patient's related haploidential donor will be divided into two portions. One portion will undergo T cell receptor (TCR) αβ depletion and the other portion will undergo CD62L depletion. Both depleted products will be infused intravenously to the patient on the same day.

ELIGIBILITY:
Inclusion Criteria:

* Patient who requires allogeneic hematopoietic stem cell transplant, has no human leukocyte antigen (HLA)-matched sibling donor but has an HLA-haploidentical donor.
* Adequate organ function to tolerate the conditioning chemotherapy and radiotherapy
* Karnofsky or Lansky performance status score ≥50

Exclusion Criteria:

* Pregnant or lactating woman
* HIV infection
* Patients for whom alternative treatment is deemed more appropriate by treating physician
* Patients who are unlikely to benefit from haploidentical hematopoietic stem cell transplantation, e.g., terminal malignancy with multiorgan failure

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Graft failure-free, GVHD-free survival | up to 1 year
  From the date of treatment start until the date of graft failure or GVHD or death from any cause, whichever comes first, assessed up to 1 year

SECONDARY OUTCOMES:
Overall survival | up to 1 year
  From the date of treatment start until the date of death from any cause, assessed up to 1 year
Proportion of patients who develop relapse among those with malignant diseases | up to 1 year
  Relapse is defined as reappearance of biopsy-proven malignant disease after complete remission
Proportion of patients who develop graft failure | up to 1 year
  Graft failure is defined as donor cells <5% in whole blood
Proportion of patients who develop infection | up to 1 year
  Any microbiologically documented infections are included
Proportion of patients who develop acute graft-versus-host disease | up to 1 year
  Acute graft-versus-host disease is defined by MAGIC criteria
Proportion of patients who develop chronic graft-versus-host disease | up to 1 year
  Chronic graft-versus-host disease is defined by NIH criteria
Proportion of patients who develop adverse events not mentioned in outcomes 4-7 | up to 1 year
  Adverse events are graded according to Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 5 (CTCAEv5)
Blood T lymphocyte count at 3 months | at 3 months
  Mean T lymphocyte count in blood among evaluable patients
Blood T lymphocyte count at 1 year | at 1 year
  Mean T lymphocyte count in blood among evaluable patients

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cheuk, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No